CLINICAL TRIAL: NCT00647699
Title: Safety and Effectiveness of the UV-X System for Corneal Collagen Cross-Linking in Eyes With Progressive Keratoconus
Brief Title: Corneal Collagen Cross-linking for Progressive Keratoconus
Acronym: CXL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UVX-002
Record Dates: First submitted 2008-03-28; First posted 2008-04-01 (Estimated); Results first posted 2016-07-07 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Progressive Keratoconus
Keywords: keratoconus; cross-linking; riboflavin; UVA light; cornea
MeSH Terms: conditions — Keratoconus; Corneal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Corneal Collagen Cross-linking (CXL) Treatment Group (Active Comparator): riboflavin ophthalmic solution and UVA irradiation
  Interventions: Drug: riboflavin ophthalmic solution; Device: UVA Irradiation
- Control Group (Sham Comparator): riboflavin ophthalmic solution without UVA irradiation.
  Interventions: Drug: riboflavin ophthalmic solution

INTERVENTIONS:
Drug: riboflavin ophthalmic solution — riboflavin 0.1% ophthalmic solution (approximately 32 drops, or 1.6 mL)
Device: UVA Irradiation — UVA light (365 nm at an irradiance of 3 mW/cm2) for 30 minutes
  Other Names: UV-X Illumination System
  Arms: Corneal Collagen Cross-linking (CXL) Treatment Group

SUMMARY:
Prospective, randomized multicenter study to determine the safety and effectiveness of performing cornea collagen cross-linking (CXL) using riboflavin and UVA light in eyes with progressive keratoconus.

DETAILED DESCRIPTION:
This was a sham controlled study for the first three months. Patients had one eye designated as the study eye and were randomized to receive one of two study treatments (CXL or sham) in their study eye. The patients were evaluated at 1, 3, 6, and 12 months. At month 3 or later patients had the option of receiving CXL treatment in both the sham and non-study eye.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of keratoconus
* Documented progression over previous 24 months
* Decreased BSCVA
* Must complete all study visits

Exclusion Criteria:

* Prior corneal surgery or Intacs
* History of delayed wound healing

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2007-12; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersh, MD, Principal Investigator — Cornea and Laser Institute
Locations (10):
- United States (10):
  - Shiley Eye Center, La Jolla, California
  - Gordon -Weiss Vision Institute, San Diego, California
  - Center for Excellence in Eye Care, Miami, Florida
  - Price Vision Group, Indianapolis, Indiana
  - Durrie Vision, Kansas City, Kansas
  - Wilmer Eye Institute at Johns Hopkins University, Baltimore, Maryland
  - Minnesota Eye Consultants, Minneapolis, Minnesota
  - Cornea & Laser Eye Institute; Hersh Vision Group, Teaneck, New Jersey
  - Edward Harkness Eye Institute at Columbia University Medical Center, New York, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York

REFERENCES:
- [Derived] Greenstein SA, Fry KL, Hersh PS. Effect of topographic cone location on outcomes of corneal collagen cross-linking for keratoconus and corneal ectasia. J Refract Surg. 2012 Jun;28(6):397-405. doi: 10.3928/1081597X-20120518-02. PMID 22692521

RESULTS

PARTICIPANT FLOW:
Groups:
- Corneal Collagen Cross-linking (CXL) Treatment Group: riboflavin ophthalmic solution and UVA irradiation (365 nm at an irradiance of 3 mW/cm2) for 30 minutes
Period: Overall Study
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group
Started | 73 | 74
Completed | 65 | 62
Not Completed | 8 | 12
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 10
  Between 18 and 65 years | 66 | 71 | 137
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 24 | 43
  Male | 54 | 50 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 31 | 36 | 67
  Unknown or Not Reported | 35 | 35 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 7 | 14
  White | 54 | 61 | 115
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Maximum Keratometry (Kmax)
Description: The primary efficacy parameter was corneal curvature, as measured by maximum keratometry (Kmax) in the study eyes. Study success was defined as a difference of ≥1 D in the mean change in Kmax from baseline to 12 months between the CXL group and control group. Keratometry was measured manually and by pentacam.
Time Frame: baseline,12 months
Population: The ITT (intent to treat) population consisted of all treated subjects, analyzed according to the treatment actually received. For the sham study eyes that received CXL treatment after baseline, the last Kmax measurement recorded prior to receiving CXL treatment was used in the analysis for later time points.
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group
Number analyzed (Participants) | 73 | 74
diopters | -1.7 (4.7) | 0.6 (2.8)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Corneal Collagen Cross-linking (CXL) Treatment Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/73 | 3/74
Other Adverse Events (participants affected / at risk) | 57/73 | 25/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corneal Collagen Cross-linking (CXL) Treatment Group (N=73) | Control Group (N=74)
ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
infectious cat bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corneal Collagen Cross-linking (CXL) Treatment Group (N=73) | Control Group (N=74)
Corneal opacity (Eye disorders) | 35 (43) | 1 (1)
Eye pain (Eye disorders) | 13 (13) | 3 (3)
Punctate keratitis (Eye disorders) | 13 (16) | 8 (8)
Corneal striae (Eye disorders) | 11 (11) | 5 (5)
Corneal epithelial defect (Eye disorders) | 10 (11) | 1 (1)
Vision blurred (Eye disorders) | 9 (12) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 7 (7) | 1 (1)
Photophobia (Eye disorders) | 6 (6) | 0 (0)
Eyelid oedema (Eye disorders) | 5 (5) | 0 (0)
Visual acuity reduced (Eye disorders) | 5 (5) | 6 (8)
Dry Eye (Eye disorders) | 4 (5) | 2 (2)
Eye irritation (Eye disorders) | 4 (4) | 1 (1)
Eye oedema (Eye disorders) | 4 (4) | 0 (0)
Anterior chamber flare (Eye disorders) | 3 (3) | 0 (0)
Corneal disorder (Eye disorders) | 3 (3) | 0 (0)
Lacrimation increased (Eye disorders) | 3 (3) | 0 (0)
Corneal oedema (Eye disorders) | 2 (2) | 0 (0)
Diplopia (Eye disorders) | 2 (2) | 1 (1)
Foreign body sensation in eye (Eye disorders) | 2 (2) | 0 (0)
Glare (Eye disorders) | 2 (2) | 1 (1)
Ocular hyperaemia (Eye disorders) | 2 (2) | 1 (1)
Visual impairment (Eye disorders) | 2 (2) | 1 (1)
Corneal scar (Eye disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site has the right to publish or communicate study results upon the earlier of: (a) publication of a multi-center publication of the Study results coordinated by Sponsor; or (b) submission of the Study data by Sponsor to the FDA; provided that the Sponsor reviews the proposed communication of results within ninety (90) days in advance of its release. Sponsor can request delay of publication or data release to allow for filing of patent application prior to the publication or release.